CLINICAL TRIAL: NCT06891586
Title: Investigation of the Relationship Between Phoenixin-14 Levels and Echocardiographic Findings in Infants of Diabetic Mothers
Brief Title: Blood Phoenixin-14 Levels and Echocardiographic Findings in Infants of Diabetic Mothers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Melek Buyukeren, Associate Professor, Konya City Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KSH_MB_2025_2
Record Dates: First submitted 2025-03-11; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Newborn Morbidity; Newborn Complication
Keywords: NEWBORN; phoenixin-14; Infants of Diabetic Mothers

STUDY DESIGN:
Intervention Model Description: The study will consist of two groups: infants of diabetic mothers and infants of healthy mothers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baby of mother diagnosed with GDM (Experimental): For participants who provide consent, residual blood samples from routine complete blood count tests performed at the 6th postnatal hour will be collected. Additionally, infants included in the study will undergo an echocardiographic evaluation by a pediatric cardiologist between postnatal days 3 and 5.
  Interventions: Diagnostic Test: echocardiographic evaluation and blood phoenixin-14 level
- healthy infants (Experimental): For consenting participants, residual blood samples from routine tests (such as complete blood count or jaundice screening) collected at the 6th hour post-birth will be gathered. Additionally, infants included in the study will undergo echocardiographic evaluation by a pediatric cardiologist between the 3rd and 5th days after birth.
  Interventions: Diagnostic Test: echocardiographic evaluation and blood phoenixin-14 level

INTERVENTIONS:
Diagnostic Test: echocardiographic evaluation and blood phoenixin-14 level — For participants who provide consent, blood samples will be collected at 6 hours postpartum. Additionally, infants included in the study will undergo an echocardiographic evaluation by a pediatric cardiologist between postnatal days 3 and 5.

SUMMARY:
In this study, the investigators hypothesize that echocardiographic pathologies observed in infants of diabetic mothers are associated with elevated serum phoenixin-14 levels.

DETAILED DESCRIPTION:
Phoenixin is a neuropeptide that has been discovered in recent years. It was first identified as a reproductive peptide in 2013. However, subsequent studies have demonstrated that phoenixin plays a regulatory role in a wide range of physiological systems, including glucose metabolism, pain perception, appetite, anxiety, and cardiovascular regulation. Phoenixin is highly expressed in various regions of the brain, including the hypothalamus, and has also been detected in circulation and peripheral tissues. Animal studies suggest that phoenixin-14 may have a direct regulatory role in the liver.

So far, two isoforms of phoenixin have been identified: phoenixin-20, which consists of a 20-amino acid peptide, and phoenixin-14, which consists of a 14-amino acid peptide. Both peptides exhibit similar functions.

Maternal diabetes is associated with significant congenital disorders, an increased risk of preterm birth, higher prenatal morbidity, and increased mortality. It can also lead to neonatal hypoglycemia and macrosomia. One of the most concerning effects is its impact on the cardiovascular system, including transient myocardial hypertrophy, which typically resolves within 2-4 weeks after birth. Additionally, it can cause disproportionate septal thickening, left ventricular outflow tract obstruction, transient hypertrophic subaortic stenosis, and heart failure.

Animal studies have shown that phoenixin-14 plays a role in myocardial repair and the regression of cardiac hypertrophy in diabetic mice. Furthermore, phoenixin-14 has been found to significantly reduce severe oxidative stress in diabetic mice.

Existing studies on phoenixin-14 in the literature have focused on adults, and there is currently no research on phoenixin-14 levels in newborns. Based on previous studies, the investigator aim is to investigate whether there is a relationship between blood phoenixin-14 levels and echocardiographic pathologies-particularly myocardial hypertrophy and interventricular septal thickness-in infants of diabetic mothers.

Between September 2023 and October 2025, mothers of infants born to diabetic mothers (study group) at Konya City Hospital will be informed about the study, and written informed consent will be obtained if they agree to participate. Similarly, during the same period, mothers of infants born to healthy mothers (control group) will be informed about the study, and written informed consent will be obtained upon their acceptance.

For participants who provide consent, residual blood samples from routine complete blood count tests performed at the 6th postnatal hour will be collected. These samples will be processed in the biochemistry laboratory, and the serum will be separated and stored at -80°C. Once the target sample size is reached, phoenixin-14 levels will be analyzed in the collected serum samples.

The cost of the kits used for phoenixin-14 testing will be covered by the researchers. The demographic and clinical characteristics of the patients, as well as prenatal and postnatal risk factors, will be recorded in a patient data collection form. Additionally, infants included in the study will undergo an echocardiographic evaluation by a pediatric cardiologist between postnatal days 3 and 5.

The study will consist of two groups: infants of diabetic mothers and infants of healthy mothers.

The investigator's study aims to investigate the relationship between phoenixin-14 levels and echocardiographic findings (intraventricular septum thickness) between the study and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Infants of diabetic mothers
* Healthy term infants

Exclusion Criteria:

* Infants whose families did not provide consent
* Infants with a syndromic appearance or congenital heart disease

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between serum phoenixin-14 levels and echocardiographic pathologies in infants of diabetic mothers. | postnatal 5 days
  Measurement Variables:
  * Serum phoenixin-14 concentration (pg/mL).
  * Presence of pathologies related to echocardiographic intraventricular septum thickness Analysis Metric: Assessment of the relationship between serum phoenixin-14 levels and echocardiographic intraventricular septum thickness.
  Data Collection Method: Serum phoenixin-14 levels will be measured using a specific immunoassay, and echocardiographic evaluations will be conducted by a pediatric cardiologist.

CONTACTS AND LOCATIONS:
Overall Officials: MELEK BUYUKEREN, Principal Investigator — Konya City Hospital
Locations (1):
- Melek Buyukeren, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Once the study is published as a scientific article, it can be shared.

REFERENCES:
- [Background] Yosten GL, Lyu RM, Hsueh AJ, Avsian-Kretchmer O, Chang JK, Tullock CW, Dun SL, Dun N, Samson WK. A novel reproductive peptide, phoenixin. J Neuroendocrinol. 2013 Feb;25(2):206-15. doi: 10.1111/j.1365-2826.2012.02381.x. PMID 22963497
- [Background] Yao B, Lv J, Du L, Zhang H, Xu Z. Phoenixin-14 protects cardiac damages in a streptozotocin-induced diabetes mice model through SIRT3. Arch Physiol Biochem. 2024 Feb;130(1):110-118. doi: 10.1080/13813455.2021.1981946. Epub 2021 Oct 7. PMID 34618648
- [Background] Yang F, Huang P, Shi L, Liu F, Tang A, Xu S. Phoenixin 14 Inhibits High-Fat Diet-Induced Non-Alcoholic Fatty Liver Disease in Experimental Mice. Drug Des Devel Ther. 2020 Sep 22;14:3865-3874. doi: 10.2147/DDDT.S258857. eCollection 2020. PMID 33061293
- [Background] Ozdemir-Kumral ZN, Sen E, Yapici HB, Atakul N, Domruk OF, Aldag Y, Sen LS, Kanpalta Mustafaoglu F, Yuksel M, Akakin D, Erzik C, Haklar G, Imeryuz N. Phoenixin 14 ameloriates pancreatic injury in streptozotocin-induced diabetic rats by alleviating oxidative burden. J Pharm Pharmacol. 2022 Nov 4;74(11):1651-1659. doi: 10.1093/jpp/rgac055. PMID 36130115
- [Background] Yuan T, Sun Z, Zhao W, Wang T, Zhang J, Niu D. Phoenixin: A Newly Discovered Peptide with Multi-Functions. Protein Pept Lett. 2017;24(6):472-475. doi: 10.2174/0929866524666170207154417. PMID 28176660
- [Background] Billert M, Kolodziejski PA, Strowski MZ, Nowak KW, Skrzypski M. Phoenixin-14 stimulates proliferation and insulin secretion in insulin producing INS-1E cells. Biochim Biophys Acta Mol Cell Res. 2019 Dec;1866(12):118533. doi: 10.1016/j.bbamcr.2019.118533. Epub 2019 Aug 15. PMID 31422055
- [Background] Wang M, Deng SP, Chen HP, Jiang DN, Tian CX, Yang W, Wu TL, Zhu CH, Zhang Y, Li GL. Phoenixin participated in regulation of food intake and growth in spotted scat, Scatophagus argus. Comp Biochem Physiol B Biochem Mol Biol. 2018 Dec;226:36-44. doi: 10.1016/j.cbpb.2018.07.007. Epub 2018 Aug 13. PMID 30114526
- [Background] Lende M, Rijhsinghani A. Gestational Diabetes: Overview with Emphasis on Medical Management. Int J Environ Res Public Health. 2020 Dec 21;17(24):9573. doi: 10.3390/ijerph17249573. PMID 33371325